CLINICAL TRIAL: NCT04826679
Title: An Open Label, Single Arm Phase II Study of Camrelizumab in Combination With Cisplatin and Nab-paclitaxel as a Novel Neoadjuvant Pre-Surgical Therapy for Resectable HNSCC
Brief Title: Neoadjuvant Camrelizumab in Combination With Cisplatin and Nab-paclitaxel in Resectable HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xuekui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-GD1-BC-HNC-II-001
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — camrelizumab; 130-nm albumin-bound paclitaxel; Cisplatin; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Camrelizumab + Cisplatin + Nab-paclitaxel
  Camrelizumab (IV), dose= 200mg , day=1 , cycle length: 21 days. Cisplatin (IV), dose=60mg/m2, day= 1, cycle length: 21 days. Nab-paclitaxel (IV), dose=260mg/m2, day= 1, cycle length: 21 days.
  Interventions: Drug: Camrelizumab, nab-paclitaxel, cisplatin

INTERVENTIONS:
Drug: Camrelizumab, nab-paclitaxel, cisplatin — Patients receive Camrelizumab IV on day 1, nab-paclitaxel IV on day 1 and cisplatin IV on day 1.
  Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: Camrelizumab and chemotherapy

SUMMARY:
This study is a single arm phase II trial including 53 patients with T2N2-3M0、T3-4N0-3M0（III-IV） head and neck squamous cell carcinoma (HNSCC) eligible for resection, who receive neo-adjvuant Camrelizumab combined with cisplatin and Nab-paclitaxel.

This proposed study will evaluate the efficacy and safety of preoperative administration of Camrelizumab combined with chemotherapy in Head and Neck Squamous Cell Carcinoma (HNSCC) who are about to undergo surgery.

DETAILED DESCRIPTION:
In this study, eligible subject will be enrolled into study arm to accept study treatment. Objective response rate will be the primary outcome measures.

ELIGIBILITY:
Inclusion Criteria：

1. Confirmed pathologic and/or cytologic diagnosis of squamous cell carcinoma of head and neck，T2N2-3M0、T3-4N0-3M0（III-IV）（AJCC 8.0）
2. Greater than or equal to 18 and less than 65 years of age at time of study entry.
3. ECOG performance status of 0 or 1.
4. Resectable or potentially resectable lesion, without distance metastasis;
5. Measurable disease as per RECIST 1.1.
6. Screening labs must meet the following criteria and must be obtained within 14 days prior to registration:
7. Adequate hepatic、cardiac、brain and renal function as demonstrated by 1) Hematology: WBC≥4000/μL、NE≥2.000/μL、HGB≥9 g/dL、PLT≥100000/μL； 2) Renal: Serum creatinine < 1.5x ULN or CrCl > 60mL/min (if using the Cockcroft-Gault formula below): 3) Hepatic: Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3 x ULN)；AST/ALT ≤ 3 x ULN and ALP≤3 x ULN；ALB≥3g / dL；
8. Ability to understand and willingness to sign an IRB approved written informed consent document. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Severe allergic reaction to any component of PD-1 monoclonal antibodies or other monoclonal antibodies.
2. Active, known or suspected autoimmune disease, including dementia and epilepsy.
3. Has had another known invasive malignancy or unresectable cancer.
4. Coagulation dysfunction: (PT > 16S, APTT > 53s, TT > 21s, FIB < 1.5g / L), bleeding tendency or thrombolysis, anticoagulation treatment.
5. Severe cardiac disease, lung dysfunction, heart function and lung function lower than grade 3 (≤3).
6. Laboratory abnormality within 7 days before enrollment.
7. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
8. Subjects with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications before enrollment.
9. Has a known history of Human Immunodeficiency Virus (HIV).
10. Has a known history of Hepatitis B (defined as HBV DNA ≥1000 cps/mL is detected) or known active Hepatitis C virus (defined as: HCV antibody positive) infection.
11. have received anti-tumor herbs within 4 weeks before randomization.
12. Pregnant or nursing women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 9 weeks
  overall response rate

SECONDARY OUTCOMES:
pCR | 9 weeks
  Pathological Complete Response
MPR | 9 weeks
  Major Pathological Response
DCR | 9 weeks
  Disease Control Rate
PFS | 2 years
  Progression-free survival
OS | 5 years
  overall survival
Adverse events graded by CTCAE v5.0 | 90 days after the first dose of study treatment
  Percentage of adverse events that are possibly, probably or definitely related to study treatment per Criteria for Adverse Events version 5 (CTCAE v5.0).

CONTACTS AND LOCATIONS:
Overall Officials: xuekui Liu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No